CLINICAL TRIAL: NCT01538849
Title: Randomized, Double-blind, Active-controlled, Multi-center Clinical Trial to Investigate the Safety, Tolerability and Efficacy of YH4808 in Patients With Reflux Esophagitis
Brief Title: Study to Investigate the Safety, Tolerability and Efficacy of YH4808 in Patients With Reflux Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YH4808-201
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Reflux Esophagitis
MeSH Terms: conditions — Esophagitis, Peptic | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- YH4808 A mg (Twice daily) (Experimental): YH4808 A mg (Twice daily, Oral administration)
  Interventions: Drug: YH4808 A mg
- YH4808 B mg (Once daily) (Experimental): YH4808 B mg (Once daily, Oral administration)
  Interventions: Drug: YH4808 B mg
- YH4808 B mg (Twice daily) (Experimental): YH4808 B mg (Twice daily, Oral administration)
  Interventions: Drug: YH4808 B mg
- YH4808 C mg (Once daily) (Experimental): YH4808 C mg (Once daily, Oral administration)
  Interventions: Drug: YH4808 C mg
- Esomeprazole 40mg (Once daily) (Active Comparator): Esomeprazole 40mg (Once daily, Oral administration)
  Interventions: Drug: Esomeprazole 40mg

INTERVENTIONS:
Drug: Esomeprazole 40mg — 1 tablet = Esomeprazole 40 mg
  Other Names: Nexium
  Arms: Esomeprazole 40mg (Once daily)
Drug: YH4808 A mg — 1 tablet = YH4808 A mg
  Other Names: Undecided
  Arms: YH4808 A mg (Twice daily)
Drug: YH4808 B mg — 1 tablet = YH4808 B mg
  Other Names: Undecided
  Arms: YH4808 B mg (Once daily); YH4808 B mg (Twice daily)
Drug: YH4808 C mg — YH4808 C mg = 2 x YH4808 B mg
  Other Names: Undecided
  Arms: YH4808 C mg (Once daily)

SUMMARY:
This study is to investigate the optimal clinical dose and administration methods of YH4808 in patients with reflux esophagitis by evaluating the safety and efficacy after YH4808 oral administration.

DETAILED DESCRIPTION:
In the result of recent meta-analysis, there was no improvement in symptoms with the first administration of PPI in about 75% of GERD patients, and symptoms were still sustained in about 50% of patients after administration of more than 3 days. Especially the nocturnal secretion of gastric acid was not effectively inhibited, and about 25% of GERD patients could not achieve the proper therapeutic effects even after PPI treatment twice daily for 4-8 weeks.

YH4808, as a selective K+- competitive acid blocker (P-CAB), is no need for activation by gastric acid since it competitively inhibits proton pump with K+. Thus, the inhibition of gastric acid secretion by YH4808 is prompt and effective. In addition, the inhibitive effect of gastric acid secretion by stimulation of histamine is proved to be more powerful than PPI (esomeprazole) and sustained in in-vitro/in-vivo model, and 24-h inhibition of gastric acid secretion and especially nocturnal inhibition of gastric acid secretion was observed to be superior to esomeprazole with repeat doses for 7 days in healthy volunteers.

Based on these nonclinical and clinical outcomes, an exploratory phase-II clinical trial is to be conducted to determine the proper treatment dose and administration method of YH48084 for GERD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who has signed on the written consent
2. Male and female aged 20 and over
3. Endoscopically verified Reflux Esophagitis classified into Los Angeles classification Grade A, B, C or D within 2 weeks before randomisation

Exclusion Criteria:

1. History or presence of upper gastrointestinal anatomic or motor disorders
2. Other exclusions apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Healing of Reflux Esophagitis (RE) Who Were "Normal(including minimal change)" at Week 4 Out of Patients Who Were Graded "A, B, C or D" at Baseline According to Los Angeles Classification | Week 4

SECONDARY OUTCOMES:
Number of Participants With Healing of Reflux Esophagitis (RE) Who Were "Normal(including minimal change)" at Week 8 Out of Patients Who Were Graded "A, B, C or D" at Baseline According to Los Angeles Classification | Week 8
Nocturnal Symptom Free Days & Symptom Free Days | Treatment Period
Sustained resolution of symptom & Time to first sustained symptom resolution | Treatment Period
Symptom Score | Treatment Period
Serum Gastrin Level | Check at Baseline(Pre-dose), 2, 4, and 8 weeks.
Global Impression of Change (Patient, Investigator) | Check at 4, and 8 weeks.
Quality of Life | Check at Baseline(Pre-dose), 4, and 8 weeks.
Epworth Sleepiness Scale | Check at Baseline(Pre-dose), 2, 4, and 8 weeks.

OTHER OUTCOMES:
Nocturnal Symptom Free Days & Symptom Free Days | Follow-up period
Sustained resolution of symptom | Follow-up period
Symptom Score | Follow-up period
Healing Rate of Reflux Esophagitis by Baseline According to Los Angeles Classification(LA Grade A~D Subgroup Analysis) | Check at Baseline, Week 4 and Week 8
Healing Rate of Reflux Esophagitis and Symptom related endpoints by H.pylori positive or negative | Treatement & Follow-up period
Adverse events, Physical examination results, ECG, Vital sign, Lab results | Treatment & Follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Myung Gyy Choi, M.D., Ph.D., Principal Investigator — Catholic Univ. Seoul St. Mary Hospital
Locations (1):
- Seoul ST.MARY'S HOSPITAL, Seoul, South Korea